CLINICAL TRIAL: NCT04805268
Title: A Single Case Study of Hypermetabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Andreas Schulze, Principal Investigator, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1000061502
Record Dates: First submitted 2021-03-03; First posted 2021-03-18 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Hypermetabolism Due to Defect in Mitochondria; Luft Disease
MeSH Terms: conditions — Hypermetabolism due to Defect in Mitochondria; Mitochondrial Myopathies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- One subject with possible Luft's disease (Experimental): 18F-FDG will be administered I.V., approximately 1 hour prior to PET/CT scan.
  Interventions: Diagnostic Test: 18F FDG PET/CT

INTERVENTIONS:
Diagnostic Test: 18F FDG PET/CT — 18F FDG PET/CT imaging (fluorine-18-fluorodeoxyglucose positron emission tomography/computed tomography).

SUMMARY:
In the Metabolic Disorder clinic at The Hospital for Sick Children, the investigators identified a male, proband with possible Luft's disease. The investigators hypothesize that Luft's disease is caused by excess or dysregulation of brown/beige fat tissue.

To address the hypothesis, the investigators would like to assess brown fat distribution and activity in this subject.

DETAILED DESCRIPTION:
The subject will undergo a fluorine-18-fluorodeoxyglucose positron emission tomography/computed tomography (18F FDG PET/CT) at the Diagnostic Imaging unit of The Hospital for Sick Children.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hypermetabolism, possible Luft's disease.

Exclusion Criteria:

* None

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Brown/beige fat tissue distribution and activity. Measurement tool- 18F FDG PET/CT (fluorine-18-fluorodeoxyglucose positron emission tomography/computed tomography) | 1 day
  Areas of 18F-FDG uptake on PET colocalizing with regions of fat will be identified on CT (-250to -10 Hounsfield Units) and quantified by Standard Uptake Value (SUV).

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Schulze, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Canada